CLINICAL TRIAL: NCT05478200
Title: Development of a Tele-Physiotherapy Tool for the Early Management of Muskuloskeletal Pain in People With Visual Impairement (TeleEDxPhysio)
Acronym: TeleEDxPhysio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escuela Universitaria de Fisioterapia de la Once (Other)
Collaborators: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Juan Andrés Martín Gonzalo, Professor, Escuela Universitaria de Fisioterapia de la Once
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2022-07-20; First posted 2022-07-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain; Visual Impairment
Keywords: therapeutical exercise; Tele-assistance plattforms; Clinical Trial
MeSH Terms: conditions — Low Back Pain; Vision Disorders | interventions — Exercise; Educational Status; Musculoskeletal Manipulations; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-directed Therapeutical Exercise and pain education program (Experimental): Patients will receive physical exercise, combined with pain education and healthy lifestyle habits: an intervention programme consisting of 3 sessions per week for 12 weeks (total of 36 sessions). Each week there will be one face-to-face session, followed by 2 home sessions, (12 face-to-face and 24 home sessions). The sessions will include cardiovascular exercises, 2 days a week we will work on strength 13 and 1 day a week we will work on mobility and exercises to improve movement control, both before the cardiovascular effort14 . Each session will include a light warm-up (at the beginning of the session) and a cool down (at the end).
  Interventions: Behavioral: physical exercise
- Pain release passive therapy based on manual therapy, thermotherapy and electroanalgesia (Active Comparator): Patients will receive 35-40 minutes of passive analgesic techniques sessions (2 per week, over 8 weeks). The following treatment will be applied:
  15 minutes of massage on the lumbopelvic musculature, lower lumbar segments and sacroiliac joints rhytmic-passive mobilization. The hip may also be mobilised at physiotherapist's discretion, 10 minutes of electrotherapy (interferential current in the lumbar region) Medium frequency current, interrupted alternating sinusoidal pulse with a frequency of up to 250 Hz and thermotherapy (10-15 minutes local in the lumbar region) with antenna electrodes placed at a distance of 20 cm from the patient's skin, at an intensity of 70 to 120 watts.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Behavioral: physical exercise — Group A (physical exercise, combined with pain education and healthy lifestyle habits), will receive an intervention programme consisting of 3 sessions per week for 12 weeks (total of 36 sessions). Each week there will be one face-to-face session, followed by 2 home sessions, (12 face-to-face and 24 home sessions). The sessions will include cardiovascular exercises, 2 days a week we will work on strength13 and 1 day a week we will work on mobility and exercises to improve movement control, both before the cardiovascular effort14 . Each session will include a light warm-up (at the beginning of the session) and a cool down (at the end).
  Other Names: education
  Arms: Semi-directed Therapeutical Exercise and pain education program
Other: Manual therapy — Group B will receive a treatment based on passive analgesic techniques consisting of manual therapy, electrotherapy (interferential currents) and thermotherapy (microwaves). This treatment will be carried out in two weekly sessions (over eight weeks) of 40 minutes each, consisting of 15 minutes of manual therapy (of the lumbopelvic musculature), 10 minutes of electrotherapy (interferential current in the lumbar region) and thermotherapy (10 minutes local in the lumbar region).
  Other Names: electrotherapy
  Arms: Pain release passive therapy based on manual therapy, thermotherapy and electroanalgesia

SUMMARY:
Chronic NonSpecific Low Back Pain (CNSLBP) is a common musculoskeletal condition often resulting in physical inactivity and disability. CNSLBP is associated with a large number of social and health costs, being one of the most important health problems worldwide. Although Therapeutical Exercise (TE) has been shown to be effective in increasing physical activity tolerance, physical fitness, strength, self perceived quality of live, pain tolerance, and overall physical activity participation levels in persons with CNSLBP, pain-release-passive therapy modalities are significantly more commonly used in clinical settings at present. On the other hand, the use of tele-assistance platforms PTAs has been gaining importance in the treatment of CNSLBP patients, especially in the use of semi-directed TE programs. However, current PTAs are not accessible for the visually impaired, a group that is at greater risk of suffering from sedentary lifestyles, restricted mobility and musculoskeletal pain due to postural or gait changes. The main hypothesis of these study is that a semi-directed TE and health education programm, in people with and without visual impairment, achieves better results in movement capacity, functional recovery, strength and compared to passive analgesic treatment in patients with CNSLBP. In a second objective, we will assess the efficacy and usability of a new PTA accesible tool for the follow-up of patients with CNSLBP who are visually impaired.

DETAILED DESCRIPTION:
INTRODUCTION Chronic non-specific low back pain (CNSLBP) is self-defining, as it is a long-lasting low back pain for which the exact cause is unknown in most cases. CLBP is a disease that causes pain and disability). It has a high social impact, as it often causes unemployment and early retirement, representing a major threat and burden to health, society and the economy. CNSLBP is associated with a high burden of direct costs, such as treatment costs (consultations, hospitalisation, medication, diagnosis, and emergency services) as well as indirect costs (lost or reduced productivity, etc. It is estimated that 5% of chronic patients consume 75% of the total cost of care for this disease and it is one of the main causes of temporary disability and permanent disability. The total number of DALYs (number of years lost due to illness, disability) associated with CNSLBP in Europe amounts to 10,731,256.71 according to the 2019 global burden of disease study, and is expected to increase, especially in Western Europe. Currently, CNSLBP is considered a health priority, which does not directly impact on the risk of death but has a high impact on quality of life.

There are a myriad of therapeutic options for the treatment of CNSLBP. Undoubtedly, those that have demonstrated the best results are all active modalities. Therapy modalities with a more passive character also have a proven analgesic efficacy, but their effect does not last over time. Studies reveal similar effects when different active therapy modalities are compared, such as walking, Pilates, abdominal exercises, analytical or functional strength exercises, stretching, among others. However, to date, we have not found a protocol that integrates the best exercises of the different modalities in the optimal workloads.

HYPOTHESIS The hypothesis put forward in this project is that a programme based on semi-directed therapeutic exercise and health education, in people with and without visual impairment, achieves better results in movement capacity, functional capacity, strength and body constitution, compared to a treatment based on passive analgesic techniques, in patients with CNSLBP.

GENERAL AND SPECIFIC OBJECTIVES The overall objective of this project is to compare the impact of a semi-directed therapeutic exercise and health education programme in CLBP patients, with and without visual impairment, compared to passive analgesic treatment.

The specific objectives to be achieved are:

1. To quantify the difference in scores on the OSWESTRY LOW BACK DISABILITY QUESTIONNAIRE (ODI), between the group of patients receiving the exercise programme (group A) and the passive analgesic treatment (group B).

   The degree of disability generated by the CLBP will be compared in both groups at the beginning and at the end of the intervention. This will allow us to create a structured recommendation on the best intervention model for the treatment of these patients.
2. Quantify what are the main differences in the movement pattern of the subjects in the active group (A) and the passive group (B).

   Significant differences, which we aim to objectify, are expected in terms of movement patterns, measured by sensors, after two opposite interventions.
3. To identify differences in the results obtained with the different intervention modalities in subjects (participants) with and without visual impairment.

   It will be interesting to identify in each of the groups whether there are differences in terms of results in subjects with and without visual impairment, thus being able to establish visual impairment as a conditioning factor in the treatment process of these patients.
4. To analyse adherence to treatment in both groups. Comparing the number of drop-outs in both groups, as well as the degree of compliance with the homework tasks (group A), would allow us to identify adherence to two totally opposite treatment modalities.
5. To find the percentage of homework completion in the active group. As this is a semi-directed exercise programme, intervention group A, part of the tasks will be carried out without the presence of the physiotherapist. It will be interesting to understand what percentage of the subjects do or do not complete the home tasks, by means of activity monitoring devices.
6. To identify difficulties in the understanding and execution of home sessions by visually impaired people. We know that even for people without visual impairment, the correct understanding of tasks at home can be extremely difficult. In this case, it will be possible to identify how the visual impairment interferes with this process by monitoring the patient on a weekly basis.
7. To find out the individual effectiveness of the exercises selected in the programme.

   There is little evidence regarding the movements selected for strength work in CLBP patients. Some authors have successfully employed whole body functional work, abdominal stabilisation exercises, extensor chain strengthening exercises, gait; however, there is still a lack of work experimenting with these exercise modalities.
8. Analyse the tools used in the study for the visually impaired user.

The patient with CNSLBP and visual impairment faces some challenges in accessing digital content. It will be important to understand whether or not the elements used are effective for this population.

All these objectives seek as a common interest the contribution of scientific evidence that supports the use of intelligent sensors in musculoskeletal pathology and that, integrated in telecare PTAs and through the use of artificial intelligence, allow the physiotherapist to be able to establish with greater precision a personalised diagnosis, as well as to serve patients as a feedback system that allows them to be an active part of their diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Suffer CNSLBP of 12 weeks or more evolution, whose pain location is mainly from T12 to the gluteal folds, with or without referred pain to the lower extremities.
* Pain that is provoked and relieved by different positions, movements and activities. In other words, mechanical behaviour.
* Low back pain whose movement behaviours have a clear association with their pain disorder.

Exclusion Criteria:

* Presence of 1 or more red flags (any sign or symptom that warns of the possible presence of a serious medical condition that may cause irreversible disability or death if not treated appropriately).
* Presence of non-specific low back pain of less than 12 weeks' duration.
* Diagnosis of specific low back pain by a physician (radicular pain, herniated disc, spondylolisthesis, stenosis, etc.), any lower limb or lumbar spine surgery within the last 3 months, pregnancy, pain without clear mechanical behaviour, active rheumatological disease, progressive neurological disease, severe cardiac or other systemic medical condition, malignant disease, acute osteoarticular trauma, fractures, infections or acute vascular problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-10-06 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Oswestry Low Back Disability Questionnaire | immediately after the intervention
  ODI: this questionnaire has been designed to give information as to how the back pain has affected the ability to manage everyday life. The patient should choose between several options on a 10 questions questionnaire.

SECONDARY OUTCOMES:
30 seconds sit to stand | immediately after the intervention
  This consists of sitting down and getting up from a chair (the same movement that we will analyse with the sensors), the maximum number of times during 30 seconds. This is a marker of general strength status.
Movement analysis with sensors | immediately after the intervention
  Ability to move during the simple gesture of getting up and sitting down five times from a chair as quickly as possible and leaning forward without bending the knees
Body build (approximate percentage of fat mass and muscle mass) | immediately after the intervention
  Bioimpedance analysis: a safe, inexpensive, accurate and non-invasive method that provides data on body composition (muscle mass, fat mass and water percentage). It consists of a very low intensity electric current that collects body tissues.

CONTACTS AND LOCATIONS:
Overall Officials: João Sousa, MSc, Principal Investigator — Escuela Universitaria de Fisioterapia de la Once
Locations (2):
- Spain (2):
  - Universidad de Zaragoza (Clínica Valdespartera y CS Seminario), Zaragoza, Aragon
  - Escuela Unviersitaria de Fisioterapia de la ONCE, Madrid

REFERENCES:
- [Background] O'Sullivan P, Caneiro JP, O'Keeffe M, O'Sullivan K. Unraveling the Complexity of Low Back Pain. J Orthop Sports Phys Ther. 2016 Nov;46(11):932-937. doi: 10.2519/jospt.2016.0609. PMID 27802794
- [Background] Wertli MM, Rasmussen-Barr E, Weiser S, Bachmann LM, Brunner F. The role of fear avoidance beliefs as a prognostic factor for outcome in patients with nonspecific low back pain: a systematic review. Spine J. 2014 May 1;14(5):816-36.e4. doi: 10.1016/j.spinee.2013.09.036. Epub 2013 Oct 18. PMID 24412032
- [Background] Jonsdottir S, Ahmed H, Tomasson K, Carter B. Factors associated with chronic and acute back pain in Wales, a cross-sectional study. BMC Musculoskelet Disord. 2019 May 15;20(1):215. doi: 10.1186/s12891-019-2477-4. PMID 31092222
- [Background] Dagenais S, Tricco AC, Haldeman S. Synthesis of recommendations for the assessment and management of low back pain from recent clinical practice guidelines. Spine J. 2010 Jun;10(6):514-29. doi: 10.1016/j.spinee.2010.03.032. PMID 20494814
- [Background] Pincus T, Burton AK, Vogel S, Field AP. A systematic review of psychological factors as predictors of chronicity/disability in prospective cohorts of low back pain. Spine (Phila Pa 1976). 2002 Mar 1;27(5):E109-20. doi: 10.1097/00007632-200203010-00017. PMID 11880847
- [Background] Farioli A, Mattioli S, Quaglieri A, Curti S, Violante FS, Coggon D. Musculoskeletal pain in Europe: the role of personal, occupational, and social risk factors. Scand J Work Environ Health. 2014 Jan;40(1):36-46. doi: 10.5271/sjweh.3381. Epub 2013 Sep 5. PMID 24009006
- [Background] Adams MA. Biomechanics of back pain. Acupunct Med. 2004 Dec;22(4):178-88. doi: 10.1136/aim.22.4.178. PMID 15628775
- [Background] Fayad F, Lefevre-Colau MM, Poiraudeau S, Fermanian J, Rannou F, Wlodyka Demaille S, Benyahya R, Revel M. [Chronicity, recurrence, and return to work in low back pain: common prognostic factors]. Ann Readapt Med Phys. 2004 May;47(4):179-89. doi: 10.1016/j.annrmp.2004.01.005. French. PMID 15130717
- [Background] Stevans JM, Delitto A, Khoja SS, Patterson CG, Smith CN, Schneider MJ, Freburger JK, Greco CM, Freel JA, Sowa GA, Wasan AD, Brennan GP, Hunter SJ, Minick KI, Wegener ST, Ephraim PL, Friedman M, Beneciuk JM, George SZ, Saper RB. Risk Factors Associated With Transition From Acute to Chronic Low Back Pain in US Patients Seeking Primary Care. JAMA Netw Open. 2021 Feb 1;4(2):e2037371. doi: 10.1001/jamanetworkopen.2020.37371. PMID 33591367
- [Background] Rahimi A, Arab AM, Nourbakhsh MR, Hosseini SM, Forghany S. Lower limb kinematics in individuals with chronic low back pain during walking. J Electromyogr Kinesiol. 2020 Apr;51:102404. doi: 10.1016/j.jelekin.2020.102404. Epub 2020 Feb 17. PMID 32120055
- [Background] O'Sullivan P. It's time for change with the management of non-specific chronic low back pain. Br J Sports Med. 2012 Mar;46(4):224-7. doi: 10.1136/bjsm.2010.081638. Epub 2011 Aug 4. No abstract available. PMID 21821612
- [Background] Kim B, Yim J. Core Stability and Hip Exercises Improve Physical Function and Activity in Patients with Non-Specific Low Back Pain: A Randomized Controlled Trial. Tohoku J Exp Med. 2020 Jul;251(3):193-206. doi: 10.1620/tjem.251.193. PMID 32669487
- [Background] Fischer SC, Calley DQ, Hollman JH. Effect of an Exercise Program That Includes Deadlifts on Low Back Pain. J Sport Rehabil. 2021 Feb 24;30(4):672-675. doi: 10.1123/jsr.2020-0324. PMID 33626500
- [Background] Tjosvoll SO, Mork PJ, Iversen VM, Rise MB, Fimland MS. Periodized resistance training for persistent non-specific low back pain: a mixed methods feasibility study. BMC Sports Sci Med Rehabil. 2020 May 8;12:30. doi: 10.1186/s13102-020-00181-0. eCollection 2020. PMID 32411374
- [Background] Suh JH, Kim H, Jung GP, Ko JY, Ryu JS. The effect of lumbar stabilization and walking exercises on chronic low back pain: A randomized controlled trial. Medicine (Baltimore). 2019 Jun;98(26):e16173. doi: 10.1097/MD.0000000000016173. PMID 31261549
- [Background] Tataryn N, Simas V, Catterall T, Furness J, Keogh JWL. Posterior-Chain Resistance Training Compared to General Exercise and Walking Programmes for the Treatment of Chronic Low Back Pain in the General Population: A Systematic Review and Meta-Analysis. Sports Med Open. 2021 Mar 8;7(1):17. doi: 10.1186/s40798-021-00306-w. PMID 33683497
- [Background] Corp N, Mansell G, Stynes S, Wynne-Jones G, Morso L, Hill JC, van der Windt DA. Evidence-based treatment recommendations for neck and low back pain across Europe: A systematic review of guidelines. Eur J Pain. 2021 Feb;25(2):275-295. doi: 10.1002/ejp.1679. Epub 2020 Nov 12. PMID 33064878
- [Background] Collins FS, Varmus H. A new initiative on precision medicine. N Engl J Med. 2015 Feb 26;372(9):793-5. doi: 10.1056/NEJMp1500523. Epub 2015 Jan 30. PMID 25635347
- [Background] Ramos JS, Dalleck LC, Tjonna AE, Beetham KS, Coombes JS. The impact of high-intensity interval training versus moderate-intensity continuous training on vascular function: a systematic review and meta-analysis. Sports Med. 2015 May;45(5):679-92. doi: 10.1007/s40279-015-0321-z. PMID 25771785
- [Background] Sahrmann S. THE HOW AND WHY OF THE MOVEMENT SYSTEM AS THE IDENTITY OF PHYSICAL THERAPY. Int J Sports Phys Ther. 2017 Nov;12(6):862-869. PMID 29158948
- [Background] Morin JB, Samozino P. Interpreting Power-Force-Velocity Profiles for Individualized and Specific Training. Int J Sports Physiol Perform. 2016 Mar;11(2):267-72. doi: 10.1123/ijspp.2015-0638. Epub 2015 Dec 17. PMID 26694658
- [Background] Garcia-Hermoso A, Cerrillo-Urbina AJ, Herrera-Valenzuela T, Cristi-Montero C, Saavedra JM, Martinez-Vizcaino V. Is high-intensity interval training more effective on improving cardiometabolic risk and aerobic capacity than other forms of exercise in overweight and obese youth? A meta-analysis. Obes Rev. 2016 Jun;17(6):531-40. doi: 10.1111/obr.12395. Epub 2016 Mar 7. PMID 26948135
- [Background] Freitas SR, Mendes B, Le Sant G, Andrade RJ, Nordez A, Milanovic Z. Can chronic stretching change the muscle-tendon mechanical properties? A review. Scand J Med Sci Sports. 2018 Mar;28(3):794-806. doi: 10.1111/sms.12957. Epub 2017 Oct 9. PMID 28801950
- [Background] Lorenzetti S, Ostermann M, Zeidler F, Zimmer P, Jentsch L, List R, Taylor WR, Schellenberg F. How to squat? Effects of various stance widths, foot placement angles and level of experience on knee, hip and trunk motion and loading. BMC Sports Sci Med Rehabil. 2018 Jul 17;10:14. doi: 10.1186/s13102-018-0103-7. eCollection 2018. PMID 30026952
- [Background] Clark DR, Lambert MI, Hunter AM. Muscle activation in the loaded free barbell squat: a brief review. J Strength Cond Res. 2012 Apr;26(4):1169-78. doi: 10.1519/JSC.0b013e31822d533d. PMID 22373894
- [Background] Calatayud J, Colado JC, Martin F, Casana J, Jakobsen MD, Andersen LL. CORE MUSCLE ACTIVITY DURING THE CLEAN AND JERK LIFT WITH BARBELL VERSUS SANDBAGS AND WATER BAGS. Int J Sports Phys Ther. 2015 Nov;10(6):803-10. PMID 26618060
- [Background] Boren K, Conrey C, Le Coguic J, Paprocki L, Voight M, Robinson TK. Electromyographic analysis of gluteus medius and gluteus maximus during rehabilitation exercises. Int J Sports Phys Ther. 2011 Sep;6(3):206-23. PMID 22034614
- [Background] Dhahbi W, Chaabene H, Chaouachi A, Padulo J, G Behm D, Cochrane J, Burnett A, Chamari K. Kinetic analysis of push-up exercises: a systematic review with practical recommendations. Sports Biomech. 2022 Jan;21(1):1-40. doi: 10.1080/14763141.2018.1512149. Epub 2018 Oct 4. PMID 30284496
- [Background] McGill SM, Cannon J, Andersen JT. Muscle activity and spine load during pulling exercises: influence of stable and labile contact surfaces and technique coaching. J Electromyogr Kinesiol. 2014 Oct;24(5):652-65. doi: 10.1016/j.jelekin.2014.06.002. Epub 2014 Jun 25. PMID 25066518
- [Background] Snarr RL, Hallmark AV, Casey JC, Esco MR. Electromyographical Comparison of a Traditional, Suspension Device, and Towel Pull-Up. J Hum Kinet. 2017 Aug 1;58:5-13. doi: 10.1515/hukin-2017-0068. eCollection 2017 Sep. PMID 28828073
- [Background] Cochrane SK, Chen SH, Fitzgerald JD, Dodson JA, Fielding RA, King AC, McDermott MM, Manini TM, Marsh AP, Newman AB, Pahor M, Tudor-Locke C, Ambrosius WT, Buford TW; LIFE Study Research Group. Association of Accelerometry-Measured Physical Activity and Cardiovascular Events in Mobility-Limited Older Adults: The LIFE (Lifestyle Interventions and Independence for Elders) Study. J Am Heart Assoc. 2017 Dec 2;6(12):e007215. doi: 10.1161/JAHA.117.007215. PMID 29197830
- [Background] Smith BE, Hendrick P, Smith TO, Bateman M, Moffatt F, Rathleff MS, Selfe J, Logan P. Should exercises be painful in the management of chronic musculoskeletal pain? A systematic review and meta-analysis. Br J Sports Med. 2017 Dec;51(23):1679-1687. doi: 10.1136/bjsports-2016-097383. Epub 2017 Jun 8. PMID 28596288
- [Background] Kahraman T, Ozcan Kahraman B, Salik Sengul Y, Kalemci O. Assessment of sit-to-stand movement in nonspecific low back pain: a comparison study for psychometric properties of field-based and laboratory-based methods. Int J Rehabil Res. 2016 Jun;39(2):165-70. doi: 10.1097/MRR.0000000000000164. PMID 27031182